CLINICAL TRIAL: NCT01995357
Title: The Influence of Base Plate Adhesive Type, Shape and Application on Degree of Leak-age - a Randomized Controlled Trial in Subjects With Ileostomy and Colostomy
Brief Title: The Influence of Baseplate Adhesive on the Degree of Leakage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP244
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Colostomy Stoma; Ileostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- First Coloplast Teast A; then Coloplast Test B (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test A; Coloplast Test B; Standard product; Training + Coloplast Test A; Training + Coloplast Test B
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product
- First Coloplast Test A; Then Standard product (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test A; Standard product; Coloplast Test B; ; Training + Coloplast Test A; Training + Coloplast Test B
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product
- First Coloplast Test B; Then Colopast Test A (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test B; Coloplast Test A; Standard product; Training + Coloplast Test B; Training + Coloplast Test A
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product
- First Coloplast Test B; Then Standard product (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test b; Standard product; Coloplast Test A; Training + Coloplast Test B; Training + Coloplast Test A
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product
- First Standard product; Then Coloplast Test A (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Standard product; Coloplast Test A; Coloplast Test B; ; Training + Coloplast Test A; Training + Coloplast Test B
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product
- First Standard Product, Then Coloplast test B (Experimental): There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Standard product; Coloplast Test B; Coloplast Test A; ; Training + Coloplast Test B; Training + Coloplast Test A
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Standard product

INTERVENTIONS:
Device: Coloplast Test A — Coloplast Test A is a newly developed ostomy appliance
Device: Coloplast Test B — Coloplast Test B is a newly developed ostomy appliance.
Device: Standard product — Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.

SUMMARY:
The influence of the baseplate adhesive type, shape and application is investigated with regard to the degree of leakage.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Have had their ileostomy/colostomy for at least 3 months
4. Have a stoma with a diameter between 15 and 36 mm
5. Be able to handle the products themselves
6. Be able to use a custom cut product
7. Normally experience faeces under the base plate at least 3 times during 2 weeks
8. Currently using SenSura 1-piece flat, open or closed bag, pre-cut or custom-cut or SenSura Mio 1-piece flat, closed bag, pre-cut or custom cut
9. Be willing to test the test products without using paste and/or ring
10. Be willing to use minimum 1 test product every second day, i.e. maximum 48 hours wear time per prod-uct
11. Be suitable for participation in the investigation
12. Be able to present a negative result of a pregnancy test - for women of childbearing age

Exclusion Criteria:

1. Are currently receiving or have within the past 2 months received radio- and/or chemotherapy
2. Are currently receiving or have within the past month received local or systemic steroid treatment in the peristomal area
3. Are pregnant or breastfeeding
4. Are participating in other interventional clinical investigations or have previously participated in this investigation
5. Use irrigation during the investigation (flush the intestines with water)
6. Are currently suffering from peristomal skin problems, i.e. bleeding and/or broken skin (assessed by the investigator/investigator representative)
7. Have a loop stoma
8. Have known hypersensitivity towards any of the test products (including adhesive remover)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- First Coloplast Teast A; Then Coloplast Test B: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test A; Coloplast Test B; Standard product; Training + Coloplast Test A; Training + Coloplast Test B
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
- First Coloplast Test A; Then Standard Product: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test A; Standard product; Coloplast Test B; ; Training + Coloplast Test A; Training + Coloplast Test B
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
- First Coloplast Test B; Then Colopast Test A: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test B; Coloplast Test A; Standard product; Training + Coloplast Test B; Training + Coloplast Test A
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
- First Coloplast Test B; Then Standard Product: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Coloplast Test b; Standard product; Coloplast Test A; Training + Coloplast Test B; Training + Coloplast Test A
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
- First Standard Product; Then Coloplast Test A: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Standard product; Coloplast Test A; Coloplast Test B; ; Training + Coloplast Test A; Training + Coloplast Test B
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
- First Standard Product, Then Coloplast Test B: There are six arms in this study. The first part of the study investigated the two test products and one comparator product. In the second part of the study the subjects test the two test products again but receive training meanwhile.
  The test sequence in this arm is:
  Standard product; Coloplast Test B; Coloplast Test A; ; Training + Coloplast Test B; Training + Coloplast Test A
  Coloplast Test A: Coloplast Test A is a newly developed ostomy appliance
  Coloplast Test B: Coloplast Test B is a newly developed ostomy appliance.
  Standard product: Standard product is the subjects usual product. Only subjects that usually use the CE-marked commercially available SenSura 1-piece flat and SenSura Mio 1-piece are included in the investigation.
Period: Period 1
Arm/Group | First Coloplast Teast A; Then Coloplast Test B | First Coloplast Test A; Then Standard Product | First Coloplast Test B; Then Colopast Test A | First Coloplast Test B; Then Standard Product | First Standard Product; Then Coloplast Test A | First Standard Product, Then Coloplast Test B
Started | 4 | 3 | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | First Coloplast Teast A; Then Coloplast Test B | First Coloplast Test A; Then Standard Product | First Coloplast Test B; Then Colopast Test A | First Coloplast Test B; Then Standard Product | First Standard Product; Then Coloplast Test A | First Standard Product, Then Coloplast Test B
Started | 4 | 3 | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | First Coloplast Teast A; Then Coloplast Test B | First Coloplast Test A; Then Standard Product | First Coloplast Test B; Then Colopast Test A | First Coloplast Test B; Then Standard Product | First Standard Product; Then Coloplast Test A | First Standard Product, Then Coloplast Test B
Started | 4 | 3 | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | First Coloplast Teast A; Then Coloplast Test B | First Coloplast Test A; Then Standard Product | First Coloplast Test B; Then Colopast Test A | First Coloplast Test B; Then Standard Product | First Standard Product; Then Coloplast Test A | First Standard Product, Then Coloplast Test B
Started | 4 | 3 | 4 (The subject who did not complete period 5, erroneously used product A when B should have been used.) | 3 | 4 | 4
Completed | 4 | 3 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | First Coloplast Teast A; Then Coloplast Test B | First Coloplast Test A; Then Standard Product | First Coloplast Test B; Then Colopast Test A | First Coloplast Test B; Then Standard Product | First Standard Product; Then Coloplast Test A | First Standard Product, Then Coloplast Test B
Started | 4 (The two discontinued subjects tested zero planned B products in period 5.) | 3 | 4 | 3 | 4 (1 subject terminated due to an adverse event. Subject counted as completed as some B products tested) | 4
Completed | 2 | 3 | 3 | 3 | 4 | 4
Not Completed | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Baseline data is summarized for all subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 19
Region of Enrollment [Number; unit: participants]
  Denmark | 22

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The primary endpoint was the degree of leakage under the baseplate, which was assessed using the three innermost rings of the 32-point leakage scale, corresponding to a total of 24 points (0 indicating no leakage and 24 indicating maximum leakage).
  Results are given separately for subjects with colostomy and ileostomy. In the ileostomy group there were no SenSura Mio participants in the standard care group.
Time Frame: 10 (- 2 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colostomy ,Test A | Colostomy, Training + Test A | Colostomy, Test B | Colostomy, Training + Test B | Colostomy, Standard Care (SenSura Mio) | Colostomy, Standard Care (SenSura) | Ileostomy, Test A | Ileostomy, Training + Test A | Ileostomy, Test B | Ileostomy, Training + Test B | Ileostomy, Standard Care (SenSura)
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 13 | 3 | 6 | 5 | 6 | 5 | 6
units on a scale | 3.6 (5.0) | 2.4 (4.2) | 5.5 (5.5) | 4.8 (5.1) | 3.7 (6.5) | 3.3 (3.2) | 9.1 (5.2) | 9.7 (5.7) | 11.5 (5.3) | 12.9 (5.6) | 8.5 (5.1)

ADVERSE EVENTS:
Time Frame: Test A + Training Test A: Pooled data of Test A during part 1 and 2 of the study. Test B + Training Test B: Pooled data of Test B during part 1 and 2 of the study. Standard Care: Data from part 1 of the study only. No Adverse Events on SenSura.
Groups:
- Test A + Training Test A: Test Product A was used both during part one of the study (Test A) and part two (Training Test A) hence adverse events are reported collectively for Test Product A.
  Consequently, Test Product A is used for two periods compared to Standard care which has been used for only one.
- Test B + Training Test B: Test Product B was used both during part one of the study (Test B) and part two (Training Test B) hence adverse events are reported collectively for Test Product B.
  Consequently, Test Product B is used for two periods compared to Standard care which has been used for only one.
- Standard Care: Standard care was used only during part one of the study. i.e. for one period only.
Arm/Group | Test A + Training Test A | Test B + Training Test B | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 8/22 | 9/22 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A + Training Test A (N=22) | Test B + Training Test B (N=22) | Standard Care (N=22)
Peristomal skin irritation/broken skin/stomal bleeding (Skin and subcutaneous tissue disorders) | 6 (8) | 9 (13) | 1 (1) — Definitely, probably or possibly related to the product. Causality not defined for 2 events with Test B + Training Test B
Cold or influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) — Not related to the product
Planned operation, non-study related (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to the product
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to the product
Diarrhea or constipation (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) — Not related to the product
Pain, leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to the product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes